CLINICAL TRIAL: NCT02610751
Title: Maternal Smoking During Pregnancy and Female Fetal Testosterone Levels
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 15-063
Record Dates: First submitted 2015-10-28; First posted 2015-11-20 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Smoking
Keywords: Maternal Smoking; Female Fetal Testosterone; Anogenital Distance; Maternal Testosterone; Maternal Cotinine
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Smoking: No interventions were applied to this group. Measurements of female fetal testosterone, maternal cotinine and testosterone levels, newborn anogenital distance, second digit to fourth digit (2D:4D) finger length ratio, newborn length and birth weight are collected.
- Non-smoking: No interventions were applied to this group. Measurements of female fetal testosterone, maternal cotinine and testosterone levels, newborn anogenital distance, second digit to fourth digit (2D:4D) finger length ratio, newborn length and birth weight are collected.

SUMMARY:
* The investigators hope their study will answer the question of whether or not fetal testosterone levels are increased in female newborns exposed to nicotine as a result of maternal smoking during pregnancy. Secondarily they plan to also evaluate maternal cotinine and testosterone levels and newborn anogenital distance, second digit to fourth digit (2D:4D) finger length ratio, newborn length and birth weight.
* The investigators hope by performing this study, they will help to uncover the effect of tobacco exposure in utero on human female fetal testosterone levels, thus improving the counseling for tobacco use in pregnancy.

DETAILED DESCRIPTION:
Epidemiological studies and laboratory research performed on animal models have revealed that the effects of maternal smoking during pregnancy go beyond the perinatal period due to the effect of nicotine on increasing fetal testosterone levels. This is of great concern as an increase fetal testosterone has been linked to impaired reproductive development and infertility in both male and female offspring, early onset of menarche in females, shorter body height, increased BMI, shortened anogenital distance and low second digit to fourth digit finger length ratio. Additionally elevated fetal testosterone levels have been associated with development of psychosocial disorders such as Autism, ADHD, antisocial behavior, conduct disorder, adult criminal behavior, and sensation seeking behavior.

Although there have been a few animal studies that have investigated the effects of maternal nicotine exposure on fetal testosterone levels with review of the epidemiologic literature on subsequent adverse implications, no known human studies have been performed to further investigate the relationship between maternal smoking during pregnancy and female fetal testosterone levels.

ELIGIBILITY:
Inclusion Criteria:

* Women, >/= 18 years old
* Current singleton pregnancy
* Recruited prior to 3rd trimester lab visit
* Known female fetus confirmed by Ultrasound, typically performed 18 to 22 weeks, or later gestational age (GA)
* Self reported smoker (of at least ½ pack per day) or non-smoker documented in electronic chart.
* Eligibility will not be limited by desired mode of delivery

Exclusion Criteria:

* Patients who successfully quit smoking at <14 weeks gestation and who have not resumed smoking during the pregnancy will be excluded from the case/control arm of study.
* Patients considered light smokers, who self report smoking less than ½ pack per day.
* Patients with Polycystic Ovarian Syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smoking and non-smoking women greater than 18 years of age with a current singleton pregnancy with known female fetus confirmed by ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Female Fetal Testosterone level | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dave Dhanraj, MD, MBA, Principal Investigator — TriHealth Inc.
Locations (2):
- United States (2):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith LM, Cloak CC, Poland RE, Torday J, Ross MG. Prenatal nicotine increases testosterone levels in the fetus and female offspring. Nicotine Tob Res. 2003 Jun;5(3):369-74. doi: 10.1080/146222031000094196. PMID 12791533
- [Background] Centers for Disease Control and Prevention (US); National Center for Chronic Disease Prevention and Health Promotion (US); Office on Smoking and Health (US). How Tobacco Smoke Causes Disease: The Biology and Behavioral Basis for Smoking-Attributable Disease: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK53017/ PMID 21452462
- [Background] Duskova M, Hruskovicova H, Simunkova K, Starka L, Parizek A. The effects of smoking on steroid metabolism and fetal programming. J Steroid Biochem Mol Biol. 2014 Jan;139:138-43. doi: 10.1016/j.jsbmb.2013.05.003. Epub 2013 May 14. PMID 23685014
- [Background] Cornelius MD, Day NL. Developmental consequences of prenatal tobacco exposure. Curr Opin Neurol. 2009 Apr;22(2):121-5. doi: 10.1097/WCO.0b013e328326f6dc. PMID 19532034
- [Background] Cornelius MD, Leech SL, Goldschmidt L, Day NL. Is prenatal tobacco exposure a risk factor for early adolescent smoking? A follow-up study. Neurotoxicol Teratol. 2005 Jul-Aug;27(4):667-76. doi: 10.1016/j.ntt.2005.05.006. PMID 16014324
- [Background] Day NL, Richardson GA, Goldschmidt L, Cornelius MD. Effects of prenatal tobacco exposure on preschoolers' behavior. J Dev Behav Pediatr. 2000 Jun;21(3):180-8. PMID 10883878
- [Background] Ernst A, Kristensen SL, Toft G, Thulstrup AM, Hakonsen LB, Olsen SF, Ramlau-Hansen CH. Maternal smoking during pregnancy and reproductive health of daughters: a follow-up study spanning two decades. Hum Reprod. 2012 Dec;27(12):3593-600. doi: 10.1093/humrep/des337. Epub 2012 Oct 2. PMID 23034153
- [Background] Barbieri RL, York CM, Cherry ML, Ryan KJ. The effects of nicotine, cotinine and anabasine on rat adrenal 11 beta-hydroxylase and 21-hydroxylase. J Steroid Biochem. 1987 Jul;28(1):25-8. doi: 10.1016/0022-4731(87)90119-1. PMID 3497305
- [Background] Matta SG, Valentine JD, Sharp BM. Nicotinic activation of CRH neurons in extrahypothalamic regions of the rat brain. Endocrine. 1997 Oct;7(2):245-53. doi: 10.1007/BF02778147. PMID 9549051
- [Background] Stroud LR, Papandonatos GD, Shenassa E, Rodriguez D, Niaura R, LeWinn KZ, Lipsitt LP, Buka SL. Prenatal glucocorticoids and maternal smoking during pregnancy independently program adult nicotine dependence in daughters: a 40-year prospective study. Biol Psychiatry. 2014 Jan 1;75(1):47-55. doi: 10.1016/j.biopsych.2013.07.024. Epub 2013 Sep 10. PMID 24034414
- [Background] Benowitz NL. Cotinine as a biomarker of environmental tobacco smoke exposure. Epidemiol Rev. 1996;18(2):188-204. doi: 10.1093/oxfordjournals.epirev.a017925. No abstract available. PMID 9021312
- [Background] Benowitz NL, Jacob P 3rd, Fong I, Gupta S. Nicotine metabolic profile in man: comparison of cigarette smoking and transdermal nicotine. J Pharmacol Exp Ther. 1994 Jan;268(1):296-303. PMID 8301571
- [Background] James WH. Potential explanation of the reported association between maternal smoking and autism. Environ Health Perspect. 2013 Feb;121(2):a42. doi: 10.1289/ehp.1206268. No abstract available. PMID 23380543
- [Background] Fowler PA, Bhattacharya S, Flannigan S, Drake AJ, O'Shaughnessy PJ. Maternal cigarette smoking and effects on androgen action in male offspring: unexpected effects on second-trimester anogenital distance. J Clin Endocrinol Metab. 2011 Sep;96(9):E1502-6. doi: 10.1210/jc.2011-1100. Epub 2011 Jul 13. PMID 21752894
- [Background] Thankamony A, Ong KK, Dunger DB, Acerini CL, Hughes IA. Anogenital distance from birth to 2 years: a population study. Environ Health Perspect. 2009 Nov;117(11):1786-90. doi: 10.1289/ehp.0900881. Epub 2009 Jul 13. PMID 20049133
- [Background] Ravnborg TL, Jensen TK, Andersson AM, Toppari J, Skakkebaek NE, Jorgensen N. Prenatal and adult exposures to smoking are associated with adverse effects on reproductive hormones, semen quality, final height and body mass index. Hum Reprod. 2011 May;26(5):1000-11. doi: 10.1093/humrep/der011. Epub 2011 Feb 18. PMID 21335416
- [Background] Rizwan S, Manning JT, Brabin BJ. Maternal smoking during pregnancy and possible effects of in utero testosterone: evidence from the 2D:4D finger length ratio. Early Hum Dev. 2007 Feb;83(2):87-90. doi: 10.1016/j.earlhumdev.2006.05.005. Epub 2006 Jun 30. PMID 16814493
- [Background] James WH. An update on the hypothesis that one cause of autism is high intrauterine levels of testosterone of maternal origin. J Theor Biol. 2014 Aug 21;355:33-9. doi: 10.1016/j.jtbi.2014.03.036. Epub 2014 Apr 1. PMID 24703983
- [Background] Kandel DB, Udry JR. Prenatal effects of maternal smoking on daughters' smoking: nicotine or testosterone exposure? Am J Public Health. 1999 Sep;89(9):1377-83. doi: 10.2105/ajph.89.9.1377. PMID 10474556
- [Background] Cornelius MD, Leech SL, Goldschmidt L, Day NL. Prenatal tobacco exposure: is it a risk factor for early tobacco experimentation? Nicotine Tob Res. 2000 Feb;2(1):45-52. doi: 10.1080/14622200050011295. PMID 11072440
- [Derived] Gordon SS, Dhanraj DN, Ganga Devaiah C, Lambers DS. A Pilot Study of Exposure to Nicotine in Human Pregnancy and Maternal and Fetal Testosterone Levels at Birth. Reprod Sci. 2022 Nov;29(11):3254-3259. doi: 10.1007/s43032-022-00967-2. Epub 2022 Jun 6. PMID 35668167